CLINICAL TRIAL: NCT02539680
Title: Joint Study on Intestinal Phosphate-TRAnsporter Expression in CKD Patients
Brief Title: Intestinal Phosphate Transporter Expression in CKD Patients
Acronym: PeTRA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficiant recruitment
Sponsor: RWTH Aachen University (Other)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14-145
Record Dates: First submitted 2015-08-25; First posted 2015-09-03 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-04

CONDITIONS: Chronic Kidney Diseases
Keywords: Phosphate transporter; CKD; duodenal biopsies
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- normal renal function (Experimental): Evaluation of the expression level of phosphate transporters at the mRNA and, if possible, on the protein level.
  Interventions: Procedure: endoscopy
- CKD stage 3-5 (not on dialysis) (Experimental): Evaluation of the expression level of phosphate transporters at the mRNA and, if possible, on the protein level.
  Interventions: Procedure: endoscopy
- on dialysis (Experimental): Evaluation of the expression level of phosphate transporters at the mRNA and, if possible, on the protein level.
  Interventions: Procedure: endoscopy

INTERVENTIONS:
Procedure: endoscopy — duodenal biopsies

SUMMARY:
The aim of the present study is to study the expression of the various phosphate transporters in patients with normal or moderately impaired renal function or in patients on dialysis. In particular, the investigators want to clarify whether NaPi-IIb expression level decreases in CKD patients, which would render it a potentially inadequate pharmaceutical target in these patients.

DETAILED DESCRIPTION:
Elevated serum phosphate is a potent predictor of death and cardiovascular events in patients with renal disease. Control of serum-phosphate to desired target ranges is insufficient in many patients with advanced chronic kidney disease (CKD), in particular dialysis patients despite dietary restrictions, optimized dialysis regimens and the use of phosphate binders. One reason why for example, phosphate binders are insufficient to control phosphate uptake in the intestine or why they even loose efficacy, is a compensatory upregulation of phosphate transporters in the gut wall.

Thus, several companies attempt to specifically interfere with intestinal phosphate transporters, in particular the NaPi-IIb transporter. However, recent Chugai data obtained in experimental CKD challenge the assumption that NaPi-IIb is the major therapeutic target in this situation. In addition to NaPi-IIb, PiT-1 and -2 also might contribute to phosphate transport.

In normal human intestinal mucosa the most prominent expression of all 3 transporters is observed in the duodenum, i.e. an area, which can easily be assessed by endoscopy.

During endoscopy a biopsy for research purposes will be obtained. Chugai will evaluate the expression level of NaPi-IIb, PiT-1, PiT-2, and villin1 at the mRNA and, if possible, the protein level.

ELIGIBILITY:
Inclusion Criteria:

* Upper endoscopy for suspected or known esophageal or gastric pathology
* Upper endoscopy for screening purposes
* Written consent to take part in the study

Exclusion Criteria:

* Food intake within 8 hours prior to the endoscopy
* Major duodenal pathology, in particular duodenitis or duodenal ulcers or tumor
* Contraindication to duodenal biopsy such as bleeding disorder
* Treatment with medication known to regulate the expression or activity of intestinal phosphate transporters (e.g. nicotinamide)
* Kidney transplant patients
* Alcohol or drug abuse
* Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study
* Participation in a parallel clinical trial
* Subjects who are in any state of dependency to the sponsor or the investigators
* Employees of the sponsor or the investigators
* Subjects who have been committed to an institution by legal or regulatory order

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Differences in the expression level of phosphate transporters in the duodenal of the populations | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schlieper, PD Dr.med., Principal Investigator — Clinic for Renal and Hypertensive Disorders, Rheumatological and Immunological Diseases (Medical Clinic II)
Locations (1):
- University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Block GA, Klassen PS, Lazarus JM, Ofsthun N, Lowrie EG, Chertow GM. Mineral metabolism, mortality, and morbidity in maintenance hemodialysis. J Am Soc Nephrol. 2004 Aug;15(8):2208-18. doi: 10.1097/01.ASN.0000133041.27682.A2. PMID 15284307
- [Background] Lee GJ, Marks J. Intestinal phosphate transport: a therapeutic target in chronic kidney disease and beyond? Pediatr Nephrol. 2015 Mar;30(3):363-71. doi: 10.1007/s00467-014-2759-x. Epub 2014 Feb 5. PMID 24496589
- [Background] Marks J, Debnam ES, Unwin RJ. The role of the gastrointestinal tract in phosphate homeostasis in health and chronic kidney disease. Curr Opin Nephrol Hypertens. 2013 Jul;22(4):481-7. doi: 10.1097/MNH.0b013e3283621310. PMID 23666413